CLINICAL TRIAL: NCT05220189
Title: A Multicenter, Single-blind, Prospective Clinical Trial to Evaluate the Clinical Performance of EarlyTect® Bladder Cancer Test in the Urine DNA for Detecting Bladder Cancer Among Hematuria Patients
Brief Title: PENK Methylation Test for Detecting Bladder Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Asan Medical Center (Other)
Collaborators: Seoul National University Hospital (Other); Korea University Anam Hospital (Other); National Cancer Center, Korea (Other Government); Pusan National University Hospital (Other); Samsung Medical Center (Other); Ajou University School of Medicine (Other); Ulsan University Hospital (Other); Chonnam National University Hospital (Other); Seoul Clinical Laboratories (Unknown); Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, In Gab Jeong, MD, Professor, Asan Medical Center
Other Study IDs: 2021-1626
Record Dates: First submitted 2022-01-07; First posted 2022-02-02 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-10

CONDITIONS: Bladder Cancer; Hematuria; Benign
Keywords: Bladder cancer; Hematuria; Methylation biomarker; EarlyTect® Bladder Cancer test; Real-time PCR (LTE-qMSP); Urine
MeSH Terms: conditions — Urinary Bladder Neoplasms; Hematuria

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Residual urine samples may be archived for further research. Clinical data and samples will be kept in a manner that preserves anonymity of the subjects, using the subject ID as the only tracking information. Specimens will be stored at Genomictree and may be used for future research.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hematuria patients aged ≥40: Device: EarlyTect Bladder Cancer test, PENK methylation assay by LTE (Linear Target Enrichment)-qMSP (quantitative methylation-specific real time PCR)
  Interventions: Diagnostic Test: EarlyTect® Bladder Cancer test

INTERVENTIONS:
Diagnostic Test: EarlyTect® Bladder Cancer test — A highly accurate and sensitive real-time PCR employing Linear Target Enrichment and Quantitative Methylation-Specific PCR (LTE-qMSP) for measuring PENK methylation in urine DNA to detect bladder cancer in hematuria patients.

SUMMARY:
The primary objective of this clinical trial is to determine the sensitivity and specificity of the EarlyTect® Bladder Cancer test for bladder cancer among patients with hematuria by comparing it to the results of cystoscopy examinations.

The second objective is to compare the clinical performance of EarlyTect® Bladder Cancer test with a NMP22 test and urine cytology test with respect to bladder cancer. By histopathological examination, lesions identified during cystoscopy will be confirmed as malignant or non-malignant by histological examination.

DETAILED DESCRIPTION:
Patients with hematuria who are scheduled for cystoscopy will be asked to collect a urine sample for EarlyTect® Bladder Cancer test and will undergo NMP22 and urine cytology tests. The participants will undergo a cystoscopy within 30 days of enrollment. For confirmation of the diagnosis and stage of the tumor, representative histopathology slides from TURBT (Transurethral Resection of Bladder Tumors) may be retrieved and examined by the central pathology laboratory.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who agree to voluntarily sign an informed consent prior to the initiation of screening
* Adults aged ≥40
* Subjects who have had gross or microscopic hematuria within the 3 months
* Subjects who had no history of bladder cancer and upper tract urothelial cancer
* Subjects who will undergo cystoscopy, NMP22 test, and urine cytology within 1 month after consent

Exclusion Criteria:

* Individuals who do not agree to voluntarily sign an informed consent prior to the initiation of screening
* Subjects aged <40 years
* Subjects with a history of bladder cancer and upper tract urothelial cancer
* Female who are currently menstruating or who have had their last menstrual period within the last 3 days
* Subjects who have undergone invasive procedures in the urinary tract system within the last 3 months
* Subjects with suspected upper urothelial cancer lesions on ultrasound or CT scan
* Subjects who have previously received pelvic radiation therapy
* Subjects who have been diagnosed with other cancers and have received or are currently receiving chemotherapy or immunotherapy within 6 months
* Subjects who require treatment for an active urinary tract infection or vaginitis
* Subjects undergoing prostate cancer treatment or requiring a prostate biopsy
* Subject has any condition which, in the opinion of the investigator should preclude participation in the study

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with hematuria
Sampling Method: Non-Probability Sample
Enrollment: 1549 (Estimated)
Dates: Start 2022-02-03 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity of the EarlyTect® Bladder Cancer test | 1 year
  Sensitivity and specificity of the EarlyTect® Bladder Cancer test for detecting bladder cancer (Stages Ta high-grade and T1-T4) in patients with hematuria compared to the cystoscopy examination, both in terms of detecting bladder cancer. The reference method is the cystoscopic procedure, and lesions will be assessed histopathologically.
  EarlyTect® Bladder Cancer test includes a measurement of PENK methylation and COL2A1 as a DNA control.
  PENK methylation in urine DNA will be assessed quantitatively by Linear Target Enrichment-coupled Quantitative Methylation-Specific PCR (LTE-qMSP) using the Real-time PCR method. The results will be dichotomized by the CT (cycle threshold) cutoff value as either positive or negative. Sensitivity = 100*(positive PENK methylation test/positive cystoscopy), Specificity = 100*(negative PENK methylation test/negative cystoscopy).

SECONDARY OUTCOMES:
The performance of the EarlyTect® Bladder Cancer test | 1 year
  The performance of the EarlyTect® Bladder Cancer test in detecting Bladder cancer in hematuria patients will be compared with those of the NMP22 and urine cytology tests.

OTHER OUTCOMES:
Comparison of clinical sensitivity and specificity to the NMP22 test | 1 year
  Comparison of clinical sensitivity and specificity to the NMP22 test
Comparison of clinical sensitivity and specificity to the urine cytology test | 1 year
  Comparison of clinical sensitivity and specificity to the urine cytology test
Sensitivity of EarlyTect® Bladder Cancer test for detecting bladder cancer with stages CIS and Ta low-grade | 1 year
  Sensitivity of EarlyTect® Bladder Cancer test for detecting bladder cancer with stages CIS and Ta low-grade
Positive predictive value (PPV) and Negative predictive value (NPV) | 1 year
  Positive predictive value and negative predictive value of EarlyTect® Bladder Cancer test for detecting bladder cancer
Evaluation of clinical sensitivity and specificity in the combination of EarlyTect® Bladder Cancer and NMP22 tests | 1 year
  Clinical sensitivity and specificity in the combination of EarlyTect® Bladder Cancer and NMP22 tests for detecting bladder cancer
Evaluation of clinical sensitivity and specificity in the combination of EarlyTect® Bladder Cancer and cytology tests | 1 year
  Clinical sensitivity and specificity in the combination of EarlyTect® Bladder Cancer and cytology tests for detecting bladder cancer
Evaluation of clinical sensitivity and specificity in the combination of EarlyTect® Bladder Cancer, NMP22, and cytology tests | 1 year
  Clinical sensitivity and specificity in the combination of EarlyTect® Bladder Cancer, NMP22, and cytology tests for detecting bladder cancer

CONTACTS AND LOCATIONS:
Overall Officials: Cheol Kwak, MD PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Asan Medical Center, Seoul, South Korea

REFERENCES:
- [Background] 1. Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018;68(6):394-424. 2. Charpentier M, Gutierrez C, Guillaudeux T, Verhoest G, Pedeux R. Noninvasive urine-based tests to diagnose or detect recurrence of bladder cancer. Cancers. 2021;13:1650. 3. Freedman ND, Silverman DT, Hollenbeck AR, Schatzkin A, Abnet CC. Association between smoking and risk of bladder cancer among men and women. JAMA 2011; 306: 737-745. 4. Kitamura H, Kakehi Y. Treatment and management of high-grade T1 bladder cancer: what should we do after second TUR? Japanese Journal of Clinical Oncology. 2015;45(4):315-322. 5. Sievert KD, Amend B, Nagele U, Schilling D, Bedke J, Horstmann M et al. Economic aspects of bladder cancer: what are the benefits and costs? World J Urol. 2009;27(3):295-300. 6. Nepple KG, O'Donnell MA. The optimal management of T1 high-grade bladder cancer. Can Urol Assoc. 2009,3(suppl4):S188-92. 7. Wakui M, Shiigai T: Urinary tract cancer screening through analysis of urinary red blood cell volume distribution. Int J Urol. 2000,7(7):248-253. 8. Yafi FA, Aprikian AG, Tanguay S, Kassouf W. Patients with microscopic and gross hematuria: practice and referral patterns among primary care physicians in a universal health care system. Con Urol Assoc J. 2011;5(2):97-101. 9. Beukers W, Kandimalla R, van Houwelingen D, Kovacic H, Chin JF, Lingsma HF et al. The use of molecular analyses in voided urine for the assessment of patients with hematuria. PLOS One. 2013;8(10):e77657. 10. Chung W, Bondaruk J, Jelinek J, Lotan Y, Liang S, Czerniak B et al: Detection of bladder cancer using novel DNA methylation biomarkers in urine sediments. Cancer Epidemiol Biomarkers Prev. 2011,20(7):1483-91. 11. Oeyen E, Hoekx L, Wachter SD, Baldewijins M, Ameye F, Mertens I. Bladder cancer diagnosis and follow-up: The current status and possible role of extracellular vesicels. Mol. Sci. 2019;20(4),821 12. Sullivan PS, Chan JB, Levin MR, Rao J. Urine cytology and adjunct markers for detection and surveillance of bladder cancer. Am J Transl Res. 2010;2(4):412-40. 13. Soria, F, Droller MJ, Lotan Y, Gontero P, D'Andrea D, Gust KM et al. An up-to-date catalog of available urinary biomarkers for the surveillance of non-muscle invasive bladder cancer. World J Urol. 2018;36:1981-95. 14. Hajdijak T. UroVysion FISH test for detecting urothelial cancers: meta-analysis of diagnostic accuracy and comparison with urinary cytology testing. Urol Oncol 2008;26(6):646-51. 15. Mbeutcha A, Lucca I, Mathieu R, Lotan Y, Shariat SF. Current status of urinary biomarkers for detection and surveillance of bladder cancer. Urol Clin N AM 2016;43:47-62 16. Chung W, Bondaruk J, Jelinek J, Lotan Y, Liang S, Czerniak B, Lssa JPJ. Detection of bladder cancer using novel DNA methylation biomarkers in urine sediments. Cancer Epidermiol Biomarkers Prev. 2011;20(7):1483-91